CLINICAL TRIAL: NCT00605735
Title: A Randomized, Parallel Group, Double-Blind, Placebo-Controlled Study to Evaluate the Clinical Efficacy and Safety of BMS-582949 Given Orally to Subjects With Rheumatoid Arthritis Having an Inadequate Response to Methotrexate
Brief Title: PoC in Rheumatoid Arthritis With Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM119-015
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Rheumatoid Arthritis, NOS
MeSH Terms: conditions — Arthritis, Rheumatoid; Pyloric Stenosis, Hypertrophic | interventions — 4-(5-(cyclopropylcarbamoyl)-2-methylphenylamino)-5-methyl-N-propylpyrrolo(1,2-f)(1,2,4)triazine-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: BMS-582949
- P1 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-582949 — Tablets, Oral, 300 mg, once daily, 12 weeks
  Other Names: P38 Inflamation
  Arms: A1
Drug: Placebo — Tablets, Oral, placebo, once daily, 12 weeks
  Arms: P1

SUMMARY:
The purpose of this study is to find out if 300 mg of BMS-582949 given once daily will be more effective than placebo after 12 weeks of treatment in subjects with rheumatoid arthritis who are also taking methotrexate

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of RA for at least 6 months
* Must be taking methotrexate for at least 3 months & on a stable dose of 7.5-30 mg weekly) for 4 weeks before dosing with study medication
* Must have at least 6 swollen and at least 8 tender joints
* CRP above upper limit of normal or ESR > 28 mm/hr
* Must wash-out (stop taking) other immunosuppressant medications to treat RA (except for methotrexate) before dosing with study medication

Exclusion Criteria:

* Any infection including TB, HIV, Hepatitis B or C
* Recent infection requiring antibiotics within 4 weeks
* History of gastrointestinal disease (such as GERD, gastrointestinal ulcers, heartburn) requiring medical or surgical treatment within 3 months
* Chronic use of proton pump inhibitors (such as Losec, Prilosec, Prevacid, Nexium), H2 blockers (such as Tagamet, Pepcid, Zantac, Axid) or antacids (such as Mylanta, Maalox)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of subjects achieving an ACR 20 at Week 12 | at Week 12

SECONDARY OUTCOMES:
Proportion of subjects achieving an ACR 20 | at each scheduled visit
Proportion of subjects schieving and ACR 50 | at each scheduled visit
Proportion of subjects schieving and ACR 70 | at each scheduled visit
Percent change from baseline to each scheduled visit in DAS28 score | at each scheduled visit
Percent change from baseline to each scheduled visit in ACR scores | at each scheduled visit
Proportion of subjects schieving a 20% change in assessment of pain, disease activity and fatigue | at each scheduled visit
Percent change from baseline to each scheduled visit in HAQ score | at each scheduled visit

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (8):
  - Desert Medical Advances, Palm Desert, California
  - Orrin M. Troum,M D, Santa Monica, California
  - G. Timothy Kelly, Md, Las Vegas, Nevada
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - The Arthritis Group, Philadelphia, Pennsylvania
  - Arthritis Clinic, Jackson, Tennessee
  - Walter F Chase Md, Austin, Texas
  - Tacoma Center For Arthritis Research Ps, Tacoma, Washington
- Argentina (3):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Ciudad Autonoma de Buenos Aire, Buenos Aires
- Czechia (3):
  - Local Institution, České Budějovice
  - Local Institution, Hradec Králové
  - Local Institution, Prague
- France (3):
  - Local Institution, Bordeaux
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Paris
- Mexico (4):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Nuevo León, Nuevo León
  - Local Institution, Culiacán, Sinaloa
- Local Institution, Cheonan, Choong Chung Nam-Do, South Korea
- Spain (3):
  - Local Institution, Madrid
  - Local Institution, Santiago de C.
  - Local Institution, Vizcaya
- Taiwan (2):
  - Local Institution, Taichung
  - Local Institution, Taoyuan District

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx